CLINICAL TRIAL: NCT03240471
Title: Cast OFF Trial: One Versus Four-five Weeks of Plaster Cast Immobilization for Non-reduced Distal Radius Fractures: A Randomized Clinical Trial - A Feasibility Trial
Brief Title: Cast OFF Trial: One Versus Four-five Weeks of Plaster Cast Immobilization
Acronym: Cast-OFF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL 59217.091.17
Record Dates: First submitted 2017-07-18; First posted 2017-08-07 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2020-10

CONDITIONS: Distal Radius Fracture
Keywords: Distal radius fracture; Conservative treatment; Patient rated outcome (PRO)
MeSH Terms: conditions — Wrist Fractures | interventions — Casts, Surgical

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One week of plaster cast (Experimental): One week of plaster cast after a non-reduced distal radius fracture.
  Interventions: Procedure: One week of plaster cast
- Control; four-five weeks of plaster cast (Other): Four-five weeks of plaster cast after a non-reduced distal radius fracture, usual care.
  Interventions: Procedure: Four-Five weeks of plaster cast

INTERVENTIONS:
Procedure: One week of plaster cast — One week of plaster cast as treatment for a non-reduced distal radius fracture.
  Arms: One week of plaster cast
Procedure: Four-Five weeks of plaster cast — Four-Five weeks of plaster cast as treatment for a non-reduced distal radius fracture.
  Arms: Control; four-five weeks of plaster cast

SUMMARY:
Distal radius fracture (DRF) is a common fracture of which the incidence appears to be increasing worldwide. On average, a total of 17% of all diagnosed fractures are DRF's.

In the Dutch guideline for DRF the treatment advice for DRF, without reduction, is treatment with plaster cast or brace for one-three weeks. Despite the advice in the guideline and despite several studies from the 90's showing that plaster cast treatment of a stable DRF for one week is safe, the usual length of plaster cast treatment for stable DRF is four-six weeks. In addition, recent studies have also shown that a long period of immobilization can lead to more post traumatic pain by increasing disuse and kinesiophobia.

This evidence suggests that the usual duration (4-6 weeks) of plaster cast treatment for DRF is unnecessary.

The aim of this feasibility study is to define whether one week of plaster cast treatment is possible and can lead to better functional results, with at least the same patient satisfaction and complications. In addition, this feasibility study will be used to define the sample size of the future RCT.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Isolated acute distal radius fracture
* Closed reduction is not performed
* Non-operative treatment with cast immobilisation
* Understanding of Dutch language

Exclusion Criteria:

* Under the age of 18 or older than 75 years
* Multiple injured patient
* Reduction is indicated/performed
* Operative treatment
* Not understanding of Dutch language

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Change in patient-rated wrist evaluation (PRWE) questionnaire score | Week 6, month 3, month 6 and month 12
  Patient rated wrist evaluation score

SECONDARY OUTCOMES:
Change in disability of the Arm, Shoulder and Hand (DASH) questionnaire score | Week 6, month 3, month 6 and month 12
  In addition to the PRWE questionnaire.
Change in Short-Form 36 questionnaire score | Week 6, month 3, month 6 and month 12
  In addition to the PRWE questionnaire.
Complications | Duration of study (12 months)
  The number of participants who experienced treatment related complications scored with a checklist.
Pain after DRF | Baseline, week 6, month 3, month 6, month 12
  Pain will be assessed by a visual analog scale (VAS). Participants rate their pain level in a scale from 0 to 10; 0 representing "no pain" and 10 representing "the worst pain imaginable".

CONTACTS AND LOCATIONS:
Overall Officials: JP Frolke, Dr., Principal Investigator — Radboud University Medical Center
Locations (3):
- Netherlands (3):
  - Rijnstate hospital, Arnhem
  - Ziekenhuis Gelderse Vallei, Ede
  - Radboudumc, Nijmegen

IPD SHARING:
Plan to Share IPD: No